CLINICAL TRIAL: NCT03984526
Title: Comparison of Effect of Atropine or Ephedrine Pretreatment for Preventing Bradycardia Under Sedation With Dexmedetomidine After Spinal Anesthesia in Elderly Patients
Brief Title: Atropine or Ephedrine Pretreatment for Preventing Bradycardia in Elderly Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, yun jeong chae, Principal Investigator, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AJIRB-MED-THE-18-343
Record Dates: First submitted 2019-06-11; First posted 2019-06-13 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Anesthesia, Spinal; Dexmedetomidine; Bradycardia
MeSH Terms: conditions — Bradycardia | interventions — Saline Solution; Atropine; Ephedrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): intravenous normal saline pretreatment
  Interventions: Drug: normal saline
- Atropine group (Experimental): intravenous atropine 0.5mg pretreatment
  Interventions: Drug: atropine 0.5mg
- Ephedrine group (Experimental): intravenous ephedrine 8mg pretreatment
  Interventions: Drug: ephedrine 8mg

INTERVENTIONS:
Drug: normal saline — intravenous normal saline pretreatment at the onset of dexmedetomidine infusion
  Arms: Control group
Drug: atropine 0.5mg — intravenous atropine 0.5mg pretreatment at the onset of dexmedetomidine infusion
  Arms: Atropine group
Drug: ephedrine 8mg — intravenous ephedrine 8mg pretreatment at the onset of dexmedetomidine infusion
  Arms: Ephedrine group

SUMMARY:
Spinal anesthesia is widely used for lower extremity surgery, and sedation is often required during surgery. For sedation, propofol, midazolam and dexmedetomidine are frequently used. Dexmedetomidine is a highly selective alpha 2 receptor agonist, and has sedating and analgesic effect. Compared with propofol and midazolam, it has little or no respiratory inhibition and hemodynamically stable. It also has the effect of reducing delirium in the elderly. Dexmedetomidine has also been reported to prolong the duration of sensory and motor blockade effects of spinal anesthesia. However, several studies have reported that administration of dexmedetomidine in spinal anesthesia increases the incidence of bradycardia.

In a study of healthy young adults, concurrent administration of atropine with dexmedetomidine in spinal anesthesia significantly reduced the frequency of bradycardia requiring treatment. However, in elderly patients, it is often reported that there is little response to atropine in bradycardia, and ephedrine is more effective in treating bradycardia than atropine in the elderly.

The investigators therefore compared ephedrine and atropine as pretreatment to reduce the incidence of bradycardia when using dexmedetomidine as a sedative in elderly patients undergoing spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Undergoing orthopedic surgery under spinal anesthesia

Exclusion Criteria:

* Contraindication for spinal anesthesia
* Atrial fibrillation, atrial flutter
* Cardiac valve disease
* Neurologic disease
* initial systolic blood pressure in operating room > 160mmHg

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 102 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
The incidence of intervention for bradycardia | for 1 hour after spinal anesthesia
  The number of treatment for bradycardia which is defined as heart rate under 50 beats per minute

SECONDARY OUTCOMES:
The incidence of intervention for hypotension | for 1 hour after spinal anesthesia
  The number of treatment for hypotension which is defined as systolic blood pressure in under 100 mmHg or systolic blood pressure under the 30% of baseline systolic blood pressure
Systolic/ mean/ diastolic blood pressure | for 1 hour after spinal anesthesia
  Systolic/ mean/ diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: yun jeong chae, Ph.D, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou universitiy school of medicine, Suwon, Gyeong-gi Do, South Korea